CLINICAL TRIAL: NCT07063186
Title: Comparing Ligation Methods During Canine Retraction Stage Using Conventional Brackets: A Randomized Controlled Trial
Brief Title: Comparing Ligation Methods During Canine Retraction Stage Using Conventional Brackets
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Sivam A/L Ramasamy, Postgraduate Orthodontic Resident, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIUM_LigationStudy
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Malocclusion; Canine Retraction
Keywords: Ligation Methods; Canine Retraction; Conventional Brackets; 3D Superimposition; Two-step Retraction; Anchorage Loss; Three-dimensional Positional Change; Canine Rotation; Canine Tipping; Canine Extrusion; Intraoral Scanners
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Elastomeric power chain on all bracket wings (Experimental): This group uses an elastomeric power chain engaged on all bracket wings
  Interventions: Other: Group A - Elastomeric power chain on all bracket wings.
- Group B - Stainless steel ligatures with elastomeric power chain placed over all bracket wings (Experimental): This group involves stainless steel ligatures used to tie in the archwire on all bracket wings, with an elastomeric power chain placed over the ligatures and engaging all four bracket wings of the maxillary canine
  Interventions: Other: Group B - Stainless steel ligatures with elastomeric power chain placed over all bracket wings.
- Group C - Elastomeric modules on mesial wings and power chain on distal wings (Experimental): In this group, elastomeric modules are placed on the mesial wings, and an elastomeric power chain is engaged on the distal wings of the maxillary canine bracket
  Interventions: Other: Group C - Elastomeric modules on mesial wings and power chain on distal wings.

INTERVENTIONS:
Other: Group A - Elastomeric power chain on all bracket wings. — Elastomeric power chain is engaged on all bracket wings
  Arms: Group A - Elastomeric power chain on all bracket wings
Other: Group B - Stainless steel ligatures with elastomeric power chain placed over all bracket wings. — Stainless steel ligatures are used to tie in the archwire on all bracket wings, with an elastomeric power chain placed over the ligatures
  Arms: Group B - Stainless steel ligatures with elastomeric power chain placed over all bracket wings
Other: Group C - Elastomeric modules on mesial wings and power chain on distal wings. — Elastomeric modules are placed on the mesial wings of each bracket, while an elastomeric power chain is engaged on the distal wings
  Arms: Group C - Elastomeric modules on mesial wings and power chain on distal wings

SUMMARY:
The goal of this Randomized Controlled Trial (RCT) is to determine the most effective way to tie the main wire to the regular orthodontic brackets during the stage of orthodontic treatment where the canines are retracted. This study is for orthodontic patients aged 16 years and older who need to have their canines retracted into spaces where other teeth have been removed.

The main questions it aims to answer are:

1. What is the effect of different ways of tying the wire to the braces on how much the maxillary canine moves back using conventional brackets?
2. How do various ways of tying the wire influence unwanted movements of the maxillary canines-specifically rotation, tipping, and extrusion?
3. What is the effect of these different tying methods on how much the back molar teeth shift forward (this is called "anchorage loss") while the maxillary canine is being pulled back?

Researchers will compare three different ways of tying the wire to the braces to see if they differ in the amount of maxillary canine retraction, three-dimensional positional changes (rotation, tipping, and extrusion), and anchorage loss of maxillary first molars:

* Group A: Uses an elastic power chain that wraps around all four parts (wings) of the brace.
* Group B: Uses thin stainless-steel wires (ligatures) to tie the brace first, then an elastic power chain is placed over these wires, also wrapping around all four parts of the brace.
* Group C: Uses small elastic rings on the two front parts (mesial wings) of the brace, and an elastic power chain on the two back parts (distal wings) of the brace.

Participants will consist of orthodontic patients aged 16 years and above from the Postgraduate Orthodontic Clinic, Kulliyyah of Dentistry, IIUM, Kuantan, who require extraction of one or both maxillary first premolars, are planned for maximum anchorage using a Nance appliance, need at least 4mm of maxillary canine retraction, and have good oral hygiene.

Participants will:

* Undergo screening and provide written informed consent for participation.
* Receive a comprehensive orthodontic examination, including photographic records, impressions, and radiographs.
* Have molar bands fitted and a Nance button fabricated and cemented, followed by dental extractions of maxillary first premolars.
* Undergo bond-up with conventional stainless-steel brackets and initial archwire placement.
* Progress through an alignment and levelling phase using progressively larger archwires, culminating in a 0.019 x 0.025-inch stainless steel archwire.
* At baseline (T0) and subsequent 4-week follow-up intervals (T1, T2, T3), have intraoral three-dimensional scans taken after archwire removal.
* Receive canine retraction using elastomeric power chains delivering a standardized 150g force. This is done as a two-step retraction, where the canine is retracted in isolation.
* Continue to receive full orthodontic treatment to completion even after the data collection period ends at T3.

DETAILED DESCRIPTION:
This Randomized Controlled Trial (RCT) aims to provide objective, quantifiable data on the effectiveness of different ligation methods during the canine retraction stage. Canine retraction is a crucial phase in fixed appliance orthodontic therapy, particularly in cases involving crowding and protrusion of maxillary anterior teeth. While numerous mechanics and materials have been developed over the years for tooth movement, the choice of ligature in conventional brackets remains a subject of debate due to observed differences in tooth movement rate, biofilm formation, friction, and force application.

A significant research gap exists in the literature regarding studies that specifically investigate the effect of different ligation methods on conventional brackets concerning anchorage loss and three-dimensional positional changes of canines. Although self-ligating brackets have gained popularity, conventional brackets remain widely used and do not always show significant improvements over conventional brackets in key treatment outcomes. Furthermore, prior studies have rarely investigated canine extrusion as a parameter during retraction with various ligation methods, which this study addresses. The study seeks to provide practitioners with objective evidence to inform their choice of ligation method, potentially improving treatment efficiency by identifying methods that facilitate optimal space closure within a given timeframe and minimize unwanted tooth movements. The use of 3D intraoral scanners and digital superimposition is prioritized for its safety, simplicity, accuracy, and patient comfort in assessing tooth movement.

1. Research Aim: To evaluate and compare the effectiveness of different ligation methods during the canine retraction using conventional orthodontic brackets in terms of amount of canine retraction, three-dimensional position change of maxillary canines and anchorage loss of maxillary first molars.

2. Objectives: i. General Objective: To identify the most effective ligation method during the canine retraction stage of orthodontic treatment using conventional brackets.

ii. Specific Objectives

1. To compare the amount of maxillary canine retraction during the retraction phase using different ligation methods.
2. To evaluate three-dimensional positional change of maxillary canines (rotation, tipping and extrusion) using different ligation methods.
3. To assess anchorage loss of maxillary first molars during canine retraction using different ligation methods.

3. Research Questions:

1. What is the effect of different ligation methods on the amount of maxillary canine retraction using conventional brackets?
2. How do various ligation methods influence the three-dimensional positional changes-specifically rotation, tipping, and extrusion-of maxillary canines during retraction?
3. What is the effect of different ligation methods on the amount of anchorage loss in the maxillary first molars during canine retraction using conventional brackets?

   4. Study Design This will be a single-centre, three-arm parallel prospective randomised controlled trial. The allocation ratio will be set at 1:1:1 for the three intervention groups. Reporting will be done based on the CONSORT 2010 Guidelines

   5. Study Groups This study will consist of three-arm parallel groups as described in Table 1. The three interventions will be randomly allocated to quadrants on the upper arch of subjects.

i. Group A - Elastomeric power chain on all bracket wings. ii. Group B - Stainless steel ligatures with elastomeric power chain placed over all bracket wings.

iii. Group C - Elastomeric modules on mesial wings and power chain on distal wings.

6. Study Population Participants will consist of patients receiving fixed appliance orthodontic treatment in IIUM, Kuantan who meet the inclusion and exclusion criteria.

i. Inclusion Criteria I. Patients aged 16 years and above. II. Patients who require extraction of one or both maxillary first premolars as part of their orthodontic treatment.

III. Patient who are planned for maximum anchorage using Nance appliance. IV. Patients who require at least 4mm of maxillary canine retraction as part of their orthodontic treatment.

V. Patients with good oral hygiene.

ii. Exclusion Criteria I. Patients with craniofacial anomalies. II. Patients with systemic or bone diseases that could affect tooth movement (e.g., osteopetrosis, osteogenesis imperfecta, Paget's disease).

III. Patients on medications that may affect tooth movement. IV. Patients with hypodontia. V. Patients with poor dental health where orthodontic treatment is not feasible.

Patients who do not fulfil all the inclusion criteria or has any one of the exclusion criteria will be excluded from the study.

7. Intervention and Treatment Protocol:

i. Pre-treatment Phase: After screening and consent, a comprehensive orthodontic examination will be performed, including intraoral and extraoral photographs, alginate impressions for stone models, and panoramic and lateral cephalometric radiographs. Molar bands and a Nance button will be fabricated and cemented before dental extractions of maxillary first premolars.

ii. Bond-Up Stage: Two weeks post-extraction, preadjusted edgewise stainless-steel brackets with MBT prescription will be bonded. Initial 0.012-inch nickel titanium alloy archwires (NiTi) will be placed and ligated with A-1 Elastomeric modules.

iii. Alignment and Levelling Phase: Patients will progress through alignment using progressively larger archwires at 4-week intervals: 0.012-inch (round) NiTi, 0.016-inch (round) NiTi, 0.018 x 0.025-inch (rectangular) NiTi, and finally 0.019 x 0.025-inch (rectangular) stainless steel (SS). The final SS archwire will remain for at least 4 weeks to ensure complete alignment and levelling.

iv. Canine Retraction Stage (Baseline T0 and Follow-ups):

* At baseline (T0), the archwire will be removed for intraoral 3D scanning. After the scan, the working archwire will be re-placed. All brackets will be ligated with elastomeric modules, except for the study canine(s).
* Canine retraction will utilize elastomeric power chains stretched to approximately twice their resting length and changed at each subsequent visit. A standardized force level of 150g will be used, measured with a calibrated force gauge.
* The study employs a two-step retraction mechanics, where the maxillary canine is retracted in isolation into the extraction space using the elastomeric power chains. This approach is preferred given that a Nance button, used for anchorage standardization, would typically become embedded during en-masse retraction.

  v. Follow-up appointments (T1, T2, T3) will occur at 4-week intervals for repeated 3D intraoral scans and power chain replacement.

  8. Data Collection and Measurement: Digital intraoral scans will be performed using a calibrated Alliedstar AS 200E intraoral scanner, with images exported in Standard Triangle Language (STL) file format.

Superimposition: Scans will be superimposed using Materialise 3-matics software (Version 13.0) by a single operator (SR). The 3D surface-to-surface matching (best-fit) method will be utilized, employing specific palatal landmarks: definite points (posterior limit of the incisive papilla, right/left lateral edges of the third palatal rugae) and a vertical line along the median palatal raphe. Elective points include medial edges of the second and third palatal rugae, which may be omitted if obstructed by the Nance button. Color-coded superimposition will be used to enhance accuracy. Superimposition will be done incrementally (T1 on T0, T2 on T1, T3 on T2) to record interval changes.

9. Randomization and Blinding: Randomization: After consent, eligible patients' quadrants will be listed in Microsoft Excel and stratified by gender. A reputable online tool (Sealed Envelope Ltd. 2019) will generate separate block randomization sequences for each gender, utilizing a fixed block size of six (two assignments for each group per block).

Allocation Concealment: Group assignments will be printed on individual sheets, folded, and sealed in opaque, sequentially numbered envelopes. An independent individual not involved in recruitment or treatment will prepare and store these envelopes. Envelopes will only be opened prior to the space closure appointment (T0).

Blinding: Due to the visible nature of the interventions, patient and clinician blinding is not possible. However, assessor blinding will be ensured by using anonymized 3D scan files, which will be renamed and recoded by an independent individual before measurements and statistical analysis by the principal investigator. Group identities will remain concealed until after statistical analysis is complete.

10. Calibration and Standardization: To ensure consistency and validity, comprehensive calibration and standardization protocols will be implemented.

Investigators: All post-graduate orthodontic residents involved in treating study patients will receive training from the Principal Investigator (SR) on ligation techniques, power chain placement, intraoral scanning, force gauge usage for standardized 150g force, two-step canine retraction mechanics, archwire sequence, and Nance button design and care. This training will be supervised by Co-Supervisor Dr. Kumeran Mohan.

Measurement Calibration: The Principal Investigator (SR) will be calibrated to a gold standard (Co-Supervisor KM) on identifying specific landmarks on 3D intraoral digital scans for measurements and superimposition. Inter-rater and intra-rater reliability will be assessed using Interclass Correlation Coefficient (ICC) on ten random 3D scans.

Equipment Calibration: The force gauge and intraoral scanner will be calibrated according to manufacturer instructions by qualified technicians prior to and routinely throughout the study.

11. Data Management and Statistical Analysis: The Principal Investigator (SR) will manage all data, which will be stored in encrypted, password-locked files to maintain confidentiality.

Statistical Analysis:

Descriptive statistics will summarize outcomes. One-way ANOVA or Kruskal-Wallis test will be used for intergroup analysis (comparing the three ligation methods).

Repeated measures ANOVA will compare changes over time within groups (T0 to T1, T1 to T2, etc.).

Paired t-tests or Wilcoxon Signed Rank test will compare outcomes between right and left quadrants.

Pearson's or Spearman's correlation may be performed to assess relationships between numerical outcomes.

If ANOVA results are significant (p<0.05), a post-hoc test such as Tukey HSD will be performed.

Intention-to-Treat (ITT) analysis will be performed to account for patient dropouts or withdrawals, utilizing the last observation carried forward (LOCF) method for missing data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years and above.
* Patients who require extraction of one or both maxillary first premolars as part of their orthodontic treatment.
* Patient who are planned for maximum anchorage using Nance appliance.
* Patients who require at least 4mm of maxillary canine retraction as part of their orthodontic treatment.
* Patients with good oral hygiene.

Exclusion Criteria:

* Patients with craniofacial anomalies.
* Patients with systemic or bone diseases that could affect tooth movement (e.g., osteopetrosis, osteogenesis imperfecta, Paget's disease).
* Patients on medications that may affect tooth movement.
* Patients with hypodontia.
* Patients with poor dental health where orthodontic treatment is not feasible.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of canine retraction (millimetres /mm) | 12 weeks
  The linear distance (mm) that the maxillary canine has moved distally from baseline (T0) to subsequent intervals will be measured

SECONDARY OUTCOMES:
Canine Rotation | 12 weeks
  The displacement of the maxillary canine in the horizontal plane will be measured in degrees (°).
Canine Tipping | 12 weeks
  The change in inclination of the maxillary canine along the vertical plane measured in degrees (°)
Canine Extrusion | 12 weeks
  Canine extrusion is the vertical displacement of the canine measured in mm
Anchorage Loss (mm) | 12 weeks
  Mesial displacement of the maxillary molars during the canine retraction will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Asst. Prof. Dr. Kumeran S/O Mohan, Study Chair — International Islamic University Malaysia
Locations (1):
- International Islamic University Malaysia, Kuantan, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Need permission from MOH Malaysia and IIUM

REFERENCES:
- [Background] Cha BK, Lee JY, Jost-Brinkmann PG, Yoshida N. Analysis of tooth movement in extraction cases using three-dimensional reverse engineering technology. Eur J Orthod. 2007 Aug;29(4):325-31. doi: 10.1093/ejo/cjm019. Epub 2007 May 19. PMID 17513876
- [Background] Cattaneo PM, Tepedino M, Hansen EB, Gram AR, Cornelis MA. Operating time for wire ligation with self-ligating and conventional brackets: A standardized in vitro study. Clin Exp Dent Res. 2022 Dec;8(6):1456-1466. doi: 10.1002/cre2.642. Epub 2022 Aug 26. PMID 36017763
- [Background] Bian C, Lyu M, Zhu M, Liu M, Xie X, Weir MD, Hack GD, Masri R, Zhang K, Bai Y, Xu HHK, Zhang N. Novel antibacterial orthodontic elastomeric ligature with oral biofilm-regulatory ability to prevent enamel demineralization. Dent Mater. 2024 Oct;40(10):1534-1545. doi: 10.1016/j.dental.2024.07.015. Epub 2024 Jul 26. PMID 39060129
- [Background] Baxi S, Tripathi AA, Bhatia V, Prasad Dubey M, Kumar P, Bagde H. Self-Ligating Bracket Systems: A Comprehensive Review. Cureus. 2023 Sep 7;15(9):e44834. doi: 10.7759/cureus.44834. eCollection 2023 Sep. PMID 37809259
- [Background] Badran SA, Al-Zaben JM, Al-Taie LM, Tbeishi H, Al-Omiri MK. Comparing patient-centered outcomes and efficiency of space closure between nickel-titanium closed-coil springs and elastomeric power chains during orthodontic treatment. Angle Orthod. 2022 Jul 1;92(4):471-477. doi: 10.2319/120721-906. PMID 35348615
- [Background] Alrehaili R, Alhujaili A, Almanjhi W, Alnami H, Alsaiyari S, Alqahtani H, Alabdan R, Baamer D, Khalil A. How Effective Are the Nance Appliance and Transpalatal Arch at Reinforcing Anchorage in Extraction Cases? Cureus. 2024 May 27;16(5):e61171. doi: 10.7759/cureus.61171. eCollection 2024 May. PMID 38933638
- [Background] Al-Haifi HAA, Ishaq RAA, Al-Hammadi MSA. Salivary pH changes under the effect of stainless steel versus elastomeric ligatures in fixed orthodontic patients: a single-center, randomized controlled clinical trial. BMC Oral Health. 2021 Oct 22;21(1):544. doi: 10.1186/s12903-021-01906-4. PMID 34686168
- [Background] Al-A'athal HS, Al-Nimri K, Alhammadi MS. Analysis of canine retraction and anchorage loss in different facial types with and without piezocision: a split-mouth-design, randomized clinical trial. Angle Orthod. 2022 Nov 1;92(6):746-754. doi: 10.2319/111921-853.1. PMID 35852456
- [Background] Al Fakir H, Carey JP, Melenka GW, Nobes DS, Heo G, Major PW. Investigation into the effects of stainless steel ligature ties on the mechanical characteristics of conventional and self-ligated brackets subjected to torque. J Orthod. 2014 Sep;41(3):188-200. doi: 10.1179/1465313314Y.0000000096. Epub 2014 Mar 4. PMID 24596162
- [Background] Abu Alhaija ES, Al Shayeb RA, Al-Khateeb S, Daher HO, Daher SO. A comparative assessment of the amount and rate of orthodontic space closure toward a healed vs recent lower premolar extraction site. Angle Orthod. 2022 Jul 1;92(4):463-470. doi: 10.2319/102921-797.1. PMID 35344007
- [Background] Abd ElMotaleb MA, El-Beialy AR, El-Sharaby FA, ElDakroury AE, Eid AA. Effectiveness of low frequency vibration on the rate of canine retraction: a randomized controlled clinical trial. Sci Rep. 2024 Apr 4;14(1):7952. doi: 10.1038/s41598-024-58268-4. PMID 38575623